CLINICAL TRIAL: NCT03703271
Title: A Prospective Randomized Multicenter Clinical Control Study of Hysteroscopic Repeat Curettage as the Primal Management of Low-risk Postmolar Gestational Trophoblastic Neoplasia
Brief Title: Study of Hysteroscopic Repeat Curettage as the First-line Treatment in Low-risk Postmolar Gestational Trophoblastic Neoplasia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Sun Yat-sen University (Other); Huazhong University of Science and Technology (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZJHGTN1212
Record Dates: First submitted 2018-10-02; First posted 2018-10-11 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Gestational Trophoblastic Neoplasia
Keywords: postmolar; Gestational Trophoblastic Neoplasia; hysteroscopic; repeat curettage; methotrexate
MeSH Terms: conditions — Gestational Trophoblastic Disease | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chemotherapy (Active Comparator): Methotrexate 0.4mg/kg·d, im ,*5d started at the first day of cycle, two weeks a cycle
  Interventions: Drug: Methotrexate
- study group (Experimental): hysteroscopic repeat curettage
  Interventions: Procedure: hysteroscopic repeat curettage

INTERVENTIONS:
Drug: Methotrexate — single-agent 5-day methotrexate, two weeks a cycle
  Other Names: Methotrexate chemotherapy
  Arms: chemotherapy
Procedure: hysteroscopic repeat curettage — Study of Hysteroscopic Repeat Curettage as the First-line Treatment in Low-risk Postmolar Gestational Trophoblastic Neoplasia
  Other Names: complete curettage
  Arms: study group

SUMMARY:
Study of hysteroscopic repeat curettage as the first-line treatment in low-risk postmolar gestational trophoblastic neoplasia compared with the MTX single drug chemotherapy

DETAILED DESCRIPTION:
Gestational trophoblastic neoplasia (GTN) is a group of malignant tumors derived from placental trophoblastic cells, most of which are secondary to hydatidiform mole, and 95% of GTN patients present low-risk gestational trophoblastic neoplasia(LR-GTN).In the 1960s and 1970s, with the in-depth study of the disease, it was found that the malignant tumor was highly sensitive to chemotherapy and had ideal tumor marker HCG to guide the treatment and follow-up. Therefore, GTN was the best malignant tumor with the overall cure rate of LR-GTN nearly 100%.MTX single-drug multi-course chemotherapy is the classic treatment of LR-GTN recommended by FIGO, but most patients can develop gastrointestinal, blood and liver toxicity during chemotherapy. In addition, the longer treatment cycle also brings a lot of discomfort to patients.

In recent years, some scholars proposed that the selection of treatment regimen of LR-GTN secondary to hydatidiform pregnancy should consider the toxic and side effects of chemotherapy, the maintenance of patients' physiological functions and quality of life.Retrospective studies abroad have shown that LR-GTN delayed chemotherapy for hydatidiform mole pregnancy only started chemotherapy for LR-GTN at a certain stage of progression, and the results did not change the prognosis of LR-GTN but reduced the rate of chemotherapy.In addition, for some patients with ultra-low risk of LR-GTN in hydatidiform pregnancy undergoing hysteroscopic repeat curettage , the rate of chemotherapy can be reduced, the related costs can be reduced and the quality of life of patients can be improved.

In this prospective, multicenter, randomized, controlled clinical study, with the routine use of a gleam of MTX single drug treatment scheme for comparison, comparing uterine cavity again emptying delay chemotherapy guided by parallel hysteroscopy surgery clinical curative effect and adverse reaction, which discuss after hydatidiform mole ultra-low dangerous GTN patients with uterine cavity emptying again guided by hysteroscopy surgery as a line of ultra low dangerous GTN patients after hydatidiform mole security and feasibility of the treatmen

ELIGIBILITY:
Inclusion Criteria:

* low-risk postmolar gestational trophoblastic neoplasia (GTN)
* World Health Organization(WHO) risk score≤4
* Age≤60 years; female, Chinese women
* Initial treatment
* Performance status: Karnofsky score≥60
* Laboratory tests: WBC≥3.5×10(9)/L, ANC≥1.5×10(9)/L, PLT≥80×10(9)/L, serum bilirubin≤ 1.5 times the upper limit of normal, transaminase≤ 1.5 times the upper limit of normal,blood urea nitrogen, Cr≤ normal
* Provide written informed consent.

Exclusion Criteria:

* Patients with unconfirmed diagnosis of GTN
* Patients with placental-site trophoblastic tumor (PSTT) or epithelioid trophoblastic tumor (ETT)
* WHO risk score ≥5分
* The diameter of a single metastatic lesion in the lung was ≥2cm
* The number of lung CT metastases was≥ 5
* With severe or uncontrolled internal disease, unable to receive chemotherapy
* Concurrently participating in other clinical trials
* Unable or unwilling to sign informed consents
* Unable or unwilling to abide by protocol

Ages: 12 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 214 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
complete remission rate in firstline treatment | 2 years
  The investigators may calculate the rate of complete response at the preliminary end point of the trail

SECONDARY OUTCOMES:
Complications of hysteroscopic repeat curettage surgery | 2 years
  The investigators may record the complications of hysteroscopic repeat curettage surgery
Severity of adverse events as assessed by the WHO | 2 years
  The investigators may record the adverse events of chemotherapy as assessed by the WHO
Overall Survival Rate (OR) | 2 years
  Overall Survival Rate of the two group patients
Ovarian functional evaluation | 2 years
  The investigators may test serum level of anti-mullerian hormone (AMH) every 6 months.
The pregnancy rate | 2 years
  To calculate the pregnancy rate in an actuarial manner using the Kaplan-Meier method at the end of the trail
Menstrual cycle resuming rate | 2 years
  The investigators record the time of menstrual cycle resuming after chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Weiguo Lv, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided